CLINICAL TRIAL: NCT07315477
Title: Characteristics of Patients Intubated for Airway Protection in the Intensive Care Unit and Timing of Tracheostomy: a Retrospective Study
Brief Title: Characteristics of Patients Intubated for Airway Protection in the Intensive Care Unit and Timing of Tracheostomy
Status: Not yet recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0269-25
Record Dates: First submitted 2025-11-20; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Airway Clearance Impairment; Intubating Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients intubated due to impending airway obstruction
  Interventions: Procedure: early tracheostomy

INTERVENTIONS:
Procedure: early tracheostomy — early tracheostomy

SUMMARY:
Every year, approximately 10-15 patients are admitted to the general intensive care unit at our institution who have been intubated for airway protection for various reasons, the main ones being soft tissue infection of the head/neck, anaphylaxis with airway edema, oral and maxillofacial/ENT surgery with airway threat, and head/neck injury with airway threat. Some patients are successfully extubated after the acute condition that caused the need for ventilation in the first place has passed, and some require tracheostomy for reasons related to the primary disease (unresolved edema, continued infectious process, need for additional invasive interventions, etc.) or for reasons related to difficulty in respiratory weaning (poor awakening, muscle weakness, development of respiratory infection, etc.).

We would like to examine whether it is possible to characterize certain parameters in the above patient population that are associated with a higher likelihood of requiring tracheostomy during hospitalization (such as age Adult). In these cases, we may consider performing the tracheostomy earlier.

ELIGIBILITY:
Inclusion Criteria: All patients aged 18-99 who were admitted to the intensive care unit from January 2012 to November 2025 and ventilated for airway protection for any reason.

-

Exclusion Criteria:Patients who did not meet the above criteria or patients for whom data was missing.

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 18-99 who were admitted to the intensive care unit from January 2012 to November 2025 and ventilated for airway protection for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Subgroup of patients with highest need for tracheostomy | 1 year
  Subgroup with highest precentage of tracheostomy

IPD SHARING:
Plan to Share IPD: No